CLINICAL TRIAL: NCT04880902
Title: Volumetric Pouch Study After Laparoscopic Sleeve Gastrectomy: Effect of the Pouch Size on Excessive Weight Loss and Weight Regain
Brief Title: Volumetric Pouch Study After Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Elkhoby, Dr, assistant lecturer of General Surgery, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01006786978123
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid
Keywords: Laparoscopic Sleeve Gastrectomy; gastric reservoir; Multi-slice computer tomography
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sleeve gastrectomy followed by volumetric assessment (Experimental)
  Interventions: Procedure: sleeve gastrectomy

INTERVENTIONS:
Procedure: sleeve gastrectomy — Laparoscopic sleeve gastrectomy had evident therapeutic effects on preexisting obesity-related comorbidities. All patients were referred for abdominal MSCT with a volumetric assessment of gastric pouch within 1 month of surgery and 1 year postoperatively

SUMMARY:
This study aimed to evaluate Laparoscopic Sleeve Gastrectomy in the treatment of morbidly obese patients pre and post-operatively after 3 months, 6 months, and 1-year follow-up and assess the volumetric changes of the gastric reservoir 1 year after LSG using multi-slice computer tomography.

ELIGIBILITY:
Inclusion Criteria:

* BMI of > 40 kg/m 2 or > 35 kg/m2 with comorbidities e.g. hypertension and type 2 DM.
* All patients failed in supervised conservative management for obesity for at least 2 years.

Exclusion Criteria:

* BMI > 60
* previous bariatric surgery
* symptomatic reflux oesophagitis disease, gastric pathology (tumor, active peptic ulcer)
* Significant psychological disorder, active alcohol or substance abuse
* severe eating disorders (bulimia)
* severe systemic disease making anesthesia or surgery prohibitively risky (American Society of Anesthesiologists (ASA) class IV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Gastric volume after surgery | 1 month
  gastric reservoir volume after performance of laparoscopic sleeve gastrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh university, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No